CLINICAL TRIAL: NCT00766480
Title: An Investigational Study of Chemoradiosensitivity Prediction With Genetic Profiling of Esophageal Biopsy for Squamous Cell Carcinoma of the Esophagus
Brief Title: Study of Tissue Samples in Predicting How Well Chemotherapy and Radiation Therapy Will Kill Cancer Cells in Patients With Squamous Cell Carcinoma of the Esophagus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toyama (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000615602; TOYAMAU-TRIEC0601
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Esophageal Cancer
Keywords: squamous cell carcinoma of the esophagus; stage IIA esophageal cancer; stage IIB esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil; Radiotherapy

ARMS (2):
- Regimen 1 (Experimental): Patients receive low-dose cisplatin IV on days 1 and 29 and low-dose fluorouracil IV on days 1-4 and 29-32. Patients also undergo concurrent radiotherapy on days 1-4 and 29-32. Patients undergo salvage surgery if needed.
  Interventions: Drug: cisplatin; Drug: fluorouracil; Radiation: radiation therapy
- Regimen 2 (Experimental): Patients receive high-dose cisplatin IV on days 1 and 29 and high-dose fluorouracil IV on days 1-4 and 29-32. Patients also undergo concurrent radiotherapy and salvage surgery as in regimen 1.
  Interventions: Drug: cisplatin; Drug: fluorouracil; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
Drug: fluorouracil — Given IV
Radiation: radiation therapy — Patients undergo radiotherapy

SUMMARY:
RATIONALE: Studying samples of tumor tissue in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This clinical trial is studying tissue samples in predicting how well chemotherapy and radiation therapy will kill cancer cells in patients with squamous cell carcinoma of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

* To search for chemoradiosensitivity-related genes using a pre-treatment biopsy sample in patients with esophageal squamous cell carcinoma treated with cisplatin, fluorouracil, and concurrent radiotherapy.
* To establish an algorithm for prediction of chemoradiosensitivity in these patients.

OUTLINE: Patients receive 1 of the following treatment regimens:

* Regimen 1: Patients receive low-dose cisplatin IV on days 1 and 29 and low-dose fluorouracil IV on days 1-4 and 29-32. Patients also undergo concurrent radiotherapy on days 1-4 and 29-32. Patients undergo salvage surgery if needed.
* Regimen 2: Patients receive high-dose cisplatin IV on days 1 and 29 and high-dose fluorouracil IV on days 1-4 and 29-32. Patients also undergo concurrent radiotherapy and salvage surgery as in regimen 1.

Pre-operative biopsy samples are analyzed by DNA microarray chip to establish an algorithm for prediction of chemoradiosensitivity.

After completion of study therapy, patients are followed at 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the thoracic esophagus

  * Stage IIA, IIB, or III (except T4) disease
  * Tumor diameter < 8 cm
* No tumor extension to the cervical esophagus or cardia of the stomach
* No multiple and different histological types of cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 4,000/mm³
* Absolute neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* AST and ALT ≤ 100 IU/L
* Total serum bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 1.2 mg/dL
* Creatinine clearance ≥ 60mL/min
* SpO_2 (room air) ≥ 95%
* Not pregnant or nursing
* No abnormal ECG findings requiring treatment
* No interstitial pneumonitis or no pulmonary fibrosis
* No severe complication (e.g., heart failure, renal failure, hepatic failure, or uncontrollable diabetes mellitus)
* No collagen disease (e.g., PSS or dermatomyositis)
* No mental disease
* No active bacterial infection
* No virus infection (i.e., HBV, HCV, PTHA, or HIV)

PRIOR CONCURRENT THERAPY:

* No prior surgery for esophageal cancer
* No prior chemotherapy
* No prior chest radiotherapy

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival
1-year local progression-free survival
3-year progression-free survival
3-year overall survival
Complete histological response

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Shimada, MD, PhD, Principal Investigator — University of Toyama
Locations (20):
- Japan (20):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kurume University School of Medicine, Kurume, Fukuoka
  - Gunma University Graduate School of Medicine, Maebashi, Gunma
  - Hiroshima City Asa Hospital, Hiroshima, Hiroshima
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kagoshima University, Kagoshima, Kagoshima-ken
  - Kyoto University Hospital, Kyoto, Kyoto
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - Graduate School of Medical Science at the University of Ryukyu, Nishiharacho, Okinawa
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Osaka
  - Kinki University School of Medicine, Sayama, Osaka
  - Osaka University Graduate School of Medicine, Suita, Osaka
  - Mita Hospital at the International University of Health and Welfare, Tokyo, Tokyo
  - Tokyo Women's Medical University, Tokyo, Tokyo
  - Toyama University Hospital, Toyama, Toyama